CLINICAL TRIAL: NCT02732587
Title: A Phase 1 Study Investigating the Interactions of AZD0530 With Alcohol in Social Drinkers
Brief Title: Investigating the Interactions of AZD0530 With Alcohol in Social Drinkers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Suchitra Krishnan-Sarin, Professor, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0602001068-2; P50AA012870 (NIH)
Record Dates: First submitted 2015-11-09; First posted 2016-04-08 (Estimated); Results first posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking | interventions — saracatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 125 mg Saracatinib (Experimental): 125 mg Saracatinib once daily for 8-11 days
  Interventions: Drug: Saracatinib

INTERVENTIONS:
Drug: Saracatinib — Subjects will receive 125 mg Saracatinib for 8-11 days followed by an alcohol interaction lab session
  Other Names: AZD0530

SUMMARY:
The purpose of this alcohol-interaction pilot study is to provide information on the effect of AZD0530 (Saracatinib) on the pharmacokinetics of alcohol and on alcohol responses, including stimulation, sedation, intoxication, body sway and physiological responses. The investigators propose to test the effects of a single dose of AZD0530 (125 mg) on alcohol related responses. This is a within subjects open label study in which the investigators plan to run 8 subjects to obtain 5 completers.

DETAILED DESCRIPTION:
The purpose of this alcohol-interaction pilot study is to provide information on the effect of AZD0530 (Saracatinib) on the pharmacokinetics of alcohol and on alcohol responses, including stimulation, sedation, intoxication, body sway and physiological responses. The investigators propose to test the effects of a single dose of AZD0530 (125 mg) on alcohol related responses. This is a within subjects open label study in which the investigators plan to run 8 subjects to obtain 5 completers.

Subjects will participate in two lab sessions, one prior to taking medication and one following 8-11 days of AZD0530. During each session, participants will receive successive doses of alcohol over a 90 min period designed to raise their blood alcohol levels to 80 mg/dl; this dose was chosen because this is close to the legal limit of intoxication and to the peak blood alcohol content (BAC) we have observed in prior research studies.Subjects will be monitored throughout the lab session and will receive a phone call two days following the 2nd lab session and a follow-up appointment one week after the 2nd lab session to assess any remaining side effects from the medication.

Once it is determined that there is no change in the pharmacokinetics of alcohol or AZD0530, as well as no difference in behavioral or cognitive responses to alcohol in the presence of AZD0530, the investigators will begin the pilot study examining the effects of two doses of AZD0530 on behavioral measures related to alcohol self-administration following a fixed dose of alcohol in alcohol abusive or dependent heavy drinkers, and compare responses to those obtained from historical controls who were treated with placebo in Study 1. Subjects will be randomized to one of two doses of AZD0530 (50 mg/day or 125 mg/day) as a between subjects factor.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 21-50
2. Able to read English at 6th grade level or higher and to complete study evaluations
3. Social drinkers consuming 1- 6 standard alcoholic drinks per week and having engaged in at least one and no more than 5 binge drinking episodes in the past year.
4. BMI 19-30

Exclusion Criteria:

1. Current DSM-V abuse or dependence criteria for alcohol, dependence criteria for other substances, other than nicotine.
2. Positive test results at any appointments after the initial intake appointment on urine drug screens conducted for opiates, cocaine, marijuana, benzodiazepines and/or barbiturates.
3. Regular use of psychoactive drugs including anxiolytics and antidepressants.
4. Psychotic or otherwise severely psychiatrically disabled.
5. Medical conditions that would contraindicate the consumption of alcohol.
6. History of neurological trauma or disease, delirium, or hallucinations, or any significant systemic illness or unstable medical condition.
7. Women who are pregnant, nursing, or refuse to use a reliable method of birth control. Urine pregnancy tests will be completed at intake and prior to administration of alcohol.
8. Subjects who report disliking spirits will be excluded because hard liquor will be provided during the alcohol administration.
9. Subjects who have taken any investigational drug and/or participated in another study which involves additive blood sampling and/or interventional measures that would be considered excessive in combination with the current protocol within 4 weeks immediately preceding admission to the treatment period.
10. Subjects who report any daily drug use during the 30 days prior to randomization for the following: anxiolytics, beta blockers, central nervous system stimulants, hypnotics, non-therapeutic doses of neuroleptics and antidepressants, drugs with psychotropic activity or drugs which cause excessive sedation.
11. Subjects who have donated blood within the past six weeks.
12. Current use (within 30 days of screening) of specific psychoactive medications (e.g., typical neuroleptics, narcotic analgesics, antiparkinsonian medications, systemic corticosteroids, or medications with significant central anticholinergic activity, etc.). Current use of warfarin.
13. Current use of the following medications (CYP3A4 substrates whose metabolism may be slowed by AZD0530): carbamazepine, colchicine, cyclosporine, disopyramide, fluticasone, quinidine, vinblastine, vincristine, nifedipine. Patients taking sildenafil, tadalafil, and vardenafil will be advised to stop taking these medications for the duration of the trial. Patients cannot take the following drugs which inhibit the CYP3A4 isoenzyme: cimetidine, cyclosporine, danazol, fluconazole, grapefruit juice, HIV protease inhibitors, itraconazole, ketoconazole, macrolides, miconazole, nefazodone, omeprazole, ritonavir, and verapamil.
14. Neutropenia defined as absolute neutrophils count of <1,500/microliter.
15. Thrombocytopenia defined as platelet count <100x103/microliter.
16. Liver function tests (AST, ALT, total bilirubin) >1.5 times upper limit of normal (ULN); serum creatinine, >2 times ULN, total bilirubin>1.5 times ULN; Serum creatinine >2.0 times ULN.
17. History of interstitial lung disease.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-03-15 (Actual); Study Completion 2016-03-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CMHC, Substance Abuse Center, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited online via craigslist.com and through local flyering
Groups:
- 125 mg Saracatinib: . Subjects participated in two inpatient alcohol administration lab sessions, a baseline session and a second session after taking 125 mg of AZD0530 for 8 outpatient days. During the outpatient drug administration phase subjects came in daily to receive their medication and at that time adverse events were assessed. Subject administration of daily medication dose was observed. The baseline session allowed participants to familiarize themselves with the procedures and provide us with a medication-free comparison for the effects of AZD0530 within the same subjects. During each lab session, subjects received six successive doses of alcohol over a 90 min period designed to raise their blood alcohol levels to 80 mg/dl.
Period: Overall Study
Arm/Group | 125 mg Saracatinib
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 125 mg Saracatinib
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (2.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Safety/Tolerability of Study Medication.
Description: Number of subjects - taking 125 mg of AZD0530 (saracatinib) over 8 days - in an alcohol drinking paradigm raising blood alcohol to 80 mg/dl who had any concerning changes in physiological or behavioral outcome measures.
Time Frame: 8 days
Measure: Number; unit: participants
Groups:
- 125 mg Saracatinib: Subjects participated in two inpatient alcohol administration lab sessions, a baseline session and a second session after taking 125 mg of AZD0530 for 8 outpatient days. During the outpatient drug administration phase subjects came in daily to receive their medication and at that time adverse events were assessed. Subject administration of daily medication dose was observed. The baseline session allowed participants to familiarize themselves with the procedures and provide us with a medication-free comparison for the effects of AZD0530 within the same subjects. During each lab session, subjects received six successive doses of alcohol over a 90 min period designed to raise their blood alcohol levels to 80 mg/dl.
Arm/Group | 125 mg Saracatinib
Number analyzed (Participants) | 5
participants | 0

ADVERSE EVENTS:
Time Frame: 5 months
Description: AE's were collected using the SAFTEE: Levine J., & Schooler N.R. (1986). SAFTEE: a technique for the systematic assessment of side effects in clinical trials. Psychopharmacology Bulletin, 22(2):343-81.
Arm/Group | 125 mg Saracatinib
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 125 mg Saracatinib (N=5)
Sleepy (General disorders) | 1 (1)
Decrease in appetite (Gastrointestinal disorders) | 1 (1)
headache (General disorders) | 1 (1)
eye twitch (right) (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes